CLINICAL TRIAL: NCT05294276
Title: Prospective Registration of Taiwan Neonatal Network (TNN)
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taiwan Society of Neonatology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202110099RINA
Record Dates: First submitted 2021-12-09; First posted 2022-03-24 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Neonatal Care
Keywords: Taiwan Neonatal Network

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention related — no intervention related

SUMMARY:
The Taiwan Neonatal Network (TNN) is an organizational structure that unites the neonatal care centers of multiple hospitals and aims to improve the quality of medical care. Countries around the world have successively established their neonatal medical care network systems to improve the quality of their neonatal care. Since the establishment of the TNN system in 2016, after five years of retrospective statistical analysis of medical records, the establishment of the TNN network system and the short-term and mid-term goals have been completed. In order to continue and improve the long-term goals and objectives of the TNN system, to improve the indicators of newborn care in Taiwan and to establish a more complete preterm infant database, it is planned to change to prospective collection, and the future preterm infant data will be registered in the TNN system. And further establish a database of various preterm infant care outcome indicators and risk factors. After statistical correction, the various preterm infant care outcome indicators among different hospitals can be regarded as the benchmark learning objects of other hospitals, and based on empirical medicine. Medical quality improvement methods have improved the quality of medical care for premature infants in Taiwan.

DETAILED DESCRIPTION:
Neonatal intensive care medicine has developed very rapidly recently, especially with the help of more advanced technology and novel treatment methods, it has achieved very good results in neonatal medicine. Despite the rapid development of neonatal intensive care medicine, death cannot be avoided with continuously updated medical equipment and treatment methods. This phenomenon is even more pronounced in the medical field of premature infants. In addition, some data can be found in different NICU settings, that is, there will be different significant results. In addition, the cost of neonatal care and medical care is extremely high, and it costs at least 10,000 yuan per day in the NICU. Since the outcome of neonatal care will be affected by the quality of medical care, and the cost of neonatal care is also high, the most important key point in neonatal care is the establishment of novel treatment methods and equipment selection. is effective and highly effective.The Taiwan Neonatal Network System (Taiwan Neonatal Network) is an organizational structure that unites the neonatal care centers of several hospitals and aims to improve the quality of their medical care. Countries around the world have successively established their neonatal medical care network systems to improve the quality of their neonatal care. Taiwan has an average of nearly 200,000 newborns every year, of which 8% to 10% are premature babies, so there are nearly 20,000 premature babies every year. In recent years, its survival rate has been significantly improved. However, premature infants are a high-risk group for complications. Among them, premature infants with a birth weight of less than 1500 grams have a higher mortality and morbidity rate. Therefore, this project is based on Improve the care of premature infants and reduce mortality and sequelae of premature infants.To achieve this goal, the mission is improving the quality and safety of medical care for newborn infants through a multidisciplinary approach of coordinated program of research, education, and quality improvement projects.

ELIGIBILITY:
Inclusion Criteria:

Any newborn with a birth weight between 401 grams and 1500 grams or a number of weeks of birth between 22 weeks plus 0 days to 29 weeks plus 6 days of live birth, if one of the above two conditions is met, it meets the preliminary acceptance criteria. Another case meets any of the following conditions:

i. Newborn born in this hospital and admitted to the hospital or ii. Newborn born in this hospital but died in the delivery room (or anywhere in this hospital) before being transferred to the intensive care unit or iii. Newborn born in the outer hospital and transferred to this hospital within 28 days of birth (the newborn has not been discharged and returned home before being transferred from the previous hospital to this hospital).

Exclusion Criteria:

Nil

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborn with a birth weight between 401 grams and 1500 grams or a number of weeks of birth between 22 weeks plus 0 days to 29 weeks plus 6 days of live birth,
Sampling Method: Probability Sample
Enrollment: 26500 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of neonatal caring: Newborn Information Registration Form | through study completion, an average of 1 year
  Newborn Information Registration Form to measure all the characteristic data, morbidities and treatments, mortality for the enrolled preterm infants
Quality of neonatal caring: CLD assessment | through study completion, an average of 1 year
  Chronic Lung Disease Assessment aim to reduce the incidence of CLD
Quality of neonatal caring: EUGR assessment | through study completion, an average of 1 year
  ExtraUterine Growth Restriction assessment aim to reduce the incidence of EUGR
Quality of neonatal caring: Hypothermia Registration Form | through study completion, an average of 1 year
  Hypothermia Registration Form aim to prevent hypothermia after birth

CONTACTS AND LOCATIONS:
Overall Officials: Po-Nien Tsao, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided